CLINICAL TRIAL: NCT05031780
Title: A Phase 2/3, Double-Blind, Randomized, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy and Safety of Mitapivat in Subjects With Sickle Cell Disease
Brief Title: A Study Evaluating the Efficacy and Safety of Mitapivat (AG-348) in Participants With Sickle Cell Disease (RISE UP)
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AG348-C-020; 2021-001674-34 (EudraCT Number)
Record Dates: First submitted 2021-07-29; First posted 2021-09-02 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — mitapivat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Phase 2: Mitapivat 50 mg BID (Experimental): Double-blind Period: Mitapivat 50 milligrams (mg) twice daily (BID) for 12 weeks.
  Interventions: Drug: Mitapivat
- Phase 2: Mitapivat 100 mg BID (Experimental): Double-blind Period: Mitapivat 100 mg BID for 12 weeks.
  Interventions: Drug: Mitapivat
- Phase 2: Placebo (Placebo Comparator): Double-blind Period: Mitapivat-matching placebo for 12 weeks.
  Interventions: Other: Mitapivat-matching placebo
- Phase 2: Open-Label Extension Period (Experimental): Participants who received mitapivat 50mg BID in the double-blind period may choose to receive mitapivat 50mg BID for 216 weeks after.
  Participants who received mitapivat 100mg BID in the double-blind period may choose to receive mitapivat 100 mg BID for 216 weeks after.
  Participants who received mitapivat-matching placebo in the double-blind period, may be randomized to receive either mitapivat 50 mg or 100 mg BID for 216 weeks after.
  Interventions: Drug: Mitapivat
- Phase 3: Mitapivat 100 mg BID (Experimental): Double-blind Period: Mitapivat 100 mg BID for 52 weeks.
  Interventions: Drug: Mitapivat
- Phase 3: Placebo (Placebo Comparator): Double-blind Period: Mitapivat-matching placebo for 52 weeks.
  Interventions: Other: Mitapivat-matching placebo
- Phase 3: Open-Label Extension Period (Experimental): Participants may choose to receive mitapivat 100 mg BID for 216 weeks after the Double-blind Period.
  Participants who received mitapivat-matching placebo in the double-blind period, may choose to receive mitapivat 100 mg BID for 216 weeks after the Double-blind Period.
  Interventions: Drug: Mitapivat

INTERVENTIONS:
Drug: Mitapivat — Mitapivat tablets
  Other Names: AG-348; Mitapivat Sulfate
  Arms: Phase 2: Mitapivat 100 mg BID; Phase 2: Mitapivat 50 mg BID; Phase 2: Open-Label Extension Period; Phase 3: Mitapivat 100 mg BID; Phase 3: Open-Label Extension Period
Other: Mitapivat-matching placebo — Placebo to match 50 mg or 100 mg tablets
  Arms: Phase 2: Placebo
Other: Mitapivat-matching placebo — Placebo to match 100 mg tablets
  Arms: Phase 3: Placebo

SUMMARY:
This clinical trial is a Phase 2/3 study that will determine the recommended dose of mitapivat and evaluate the efficacy and safety of mitapivat in sickle cell disease by testing how well mitapivat works compared to placebo to increase the amount of hemoglobin in the blood and to reduce or prevent the occurrence of sickle cell pain crises. In addition, the long-term effect of mitapivat on efficacy and safety will be explored in an open-label extension portion.

DETAILED DESCRIPTION:
Mitapivat is a small molecule, oral activator of pyruvate kinase R (PKR). PKR is involved with maintaining health, energy, and longevity of red blood cells (RBCs). The study aims to evaluate the efficacy and safety of treatment with mitapivat in participants with sickle cell disease. The study is a Phase 2/3 study in which the recommended dose of mitapivat will be selected and further evaluated. The Phase 2 portion includes a 12-week randomized, placebo-controlled period in which participants will be randomized in a 1:1:1 ratio to receive 2 dose levels of mitapivat or placebo. The Phase 3 portion includes a 52-week randomized, placebo-controlled period in which participants will be randomized in a 2:1 ratio to receive the recommended mitapivat dose level or placebo. Participants who complete either the Phase 2 or Phase 3 portion will have the option to move into a 216-week open label extension period to receive mitapivat.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 years or older (18 years or older [France and Germany]); participants age 16 or 17 years must physically have completed puberty;
* Documented diagnosis of sickle cell disease (SCD) (HbSS, HbSC [combined heterozygosity for hemoglobins S and C], HbS/beta 0- thalassemia, HbS/ beta plus thalassemia, or other sickle cell syndrome variants);
* At least 2 SCPCs and no more than 10 SCPCs in the past 12 months;
* Hemoglobin at least 5.5 and 10.5 gram per deciliter (g/dL) at the most. Hemoglobin concentration must be based on an average of at least 2 Hb concentration measurements (separated by ≥7 days) collected during the Screening Period;
* If taking hydroxyurea, the hydroxyurea dose must be stable for at least 90 days before starting study drug. Discontinuation of hydroxyurea requires a 90-day washout prior to informed assent/consent;
* Women capable of becoming pregnant must agree to use 2 forms of contraception.

Exclusion Criteria:

* Pregnant, breastfeeding, or parturient;
* Receiving regularly scheduled transfusions;
* Hepatobiliary disorders including but not limited to significant liver disease or gallbladder disease;
* Severe kidney disease;
* Prior exposure to gene therapy or prior bone marrow or stem cell transplantation;
* Currently receiving treatment with a disease-modifying therapy for SCD (eg, voxelotor, crizanlizumab, L-glutamine), with the exception of hydroxyurea. The last dose of voxelotor, crizanlizumab, and L-glutamine must have been administered at least 90 days before randomization;
* Currently receiving treatment with hematopoietic stimulating agents; the last dose must have been administered at least 90 days before starting study drug;
* Received treatment on another investigational trial within 90 days prior to start of study drug or plans to participate in another investigational drug trial;
* Taking medications that are strong inhibitors of CYP3A4/5 or strong inducers of CYP3A4 that cannot be stopped in an acceptable timeframe before starting study drug (timeframe will be discussed with your doctor).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Phase 2: Percentage of Participants With Hemoglobin (Hb) Response | Week 12
Phase 2: Percentage of Participants With Treatment-Emergent Adverse Events (AEs) and Treatment-Emergent Serious AEs (SAEs) | Up to Week 12
Phase 3: Percentage of Participants With Hb Response | Week 52
Phase 3: Annualized Rate of Sickle Cell Pain Crises (SCPCs) | Up to Week 52

SECONDARY OUTCOMES:
Phase 2: Change From Baseline in Hb Concentration | Baseline, Week 10 up to Week 12
Phase 2: Change From Baseline in Indirect Bilirubin | Baseline, Week 10 up to Week 12
Phase 2: Change From Baseline in Lactate Dehydrogenase (LDH) | Baseline, Week 10 up to Week 12
Phase 2: Change From Baseline in Absolute Reticulocytes Count | Baseline, Week 10 up to Week 12
Phase 2: Change From Baseline in Percent Reticulocytes | Baseline, Week 10 up to Week 12
Phase 2: Change From Baseline in Erythropoietin | Baseline, Week 10 up to Week 12
Phase 2: Change From Baseline in Patient-Reported Outcomes Measurement Information System® (PROMIS®) Fatigue 13a Short Form (SF) Score | Baseline, Week 10 up to Week 12
Phase 2: Annualized Rate of SCPCs | Up to Week 12
Phase 2: Pharmacokinetic/Pharmacodynamic Relationship: Evaluate the Exposure of Mitapivat to the Change in Adenosine Triphosphate (ATP) and 2,3-Diphosphoglycerate (2,3-DPG) | Day 1 up to Week 8
Phase 2: Mitapivat Concentration Over Time | Day 1 up to Week 8
Phase 2: Mitapivat Area Under the Concentration | Day 1 up to Week 8
Phase 2: Mitapivat Maximum (Peak) Concentration | Day 1 up to Week 8
Phase 3: Change From Baseline in Hb Concentration | Baseline, Week 24 up to Week 52
Phase 3: Change From Baseline in Indirect Bilirubin | Baseline, Week 24 up to Week 52
Phase 3: Change From Baseline in Percent Reticulocytes | Baseline, Week 24 up to Week 52
Phase 3: Change From Baseline in PROMIS® Fatigue 13a SF Scores | Baseline, Week 24 up to Week 52
Phase 3: Annualized Frequency of Hospitalizations for SCPC | Up to Week 52
Phase 3: Change From Baseline in LDH Concentration | Baseline, Week 24 up to Week 52
Phase 3: Change From Baseline in Absolute Reticulocytes | Baseline, Week 24 up to Week 52
Phase 3: Change From Baseline in Erythropoietin | Baseline, Week 24 up to Week 52
Phase 3: Percentage of Participants With Improvement in the Patient Global Impression of Severity (PGIS) -Fatigue | Baseline, Weeks 24, 28, 40, and 52
Phase 3: Percentage of Participants With Improvement in the Patient Global Impression of Change (PGIC) -Fatigue | Baseline, Weeks 24, 28, 40, and 52
Phase 3: Time to First SCPC | Up to Week 52
Phase 3: Time to Second SCPC | Up to Week 52
Phase 3: Annualized Rate of Hospitalization Days for SCPC | Up to Week 52
Phase 3: Annualized Rate of Emergency Room Visits for SCPC | Up to Week 52
Phase 3: Change From Baseline in 6-Minute Walk Test (6MWT) | Baseline, Week 52
Phase 3: Change From Baseline in PROMIS Pain Intensity | Baseline, Week 24 and 52
Phase 3: Change From Baseline in Adult Sickle Cell Quality of Life Measurement Information System (ASCQ-Me) Pain Impact | Baseline, Week 24 and 52
Phase 3: PGIC of Pain | Baseline, Week 52
Phase 3: Change From Baseline in PGIS of Pain | Baseline, Week 52
Phase 3: Percentage of Participants With Treatment-Emergent Adverse Events (AEs) and Treatment-Emergent Serious AEs (SAEs) | Up to 56 weeks
Phase 3: Pharmacokinetic/Pharmacodynamic Relationship: Evaluate the Exposure of Mitapivat to the Change in ATP and 2,3-DPG Levels | Day 1 up to Week 40
Phase 3: Mitapivat Concentration Over Time | Day 1 up to Week 40
Phase 3: Mitapivat Area Under the Concentration Curve | Day 1 up to Week 40
Phase 3: Mitapivat Maximum (Peak) Concentration | Day 1 up to Week 40

CONTACTS AND LOCATIONS:
Locations (90):
- United States (28):
  - University of California San Diego, La Jolla, California
  - UCLA Health, Los Angeles, California
  - Children's Hospital Oakland, Oakland, California
  - University of Connecticut Health Center, Farmington, Connecticut
  - Children's National Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Sylvester Comprehensive Cancer Center-Miami, Miami, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Riley Hospital For Children, Indianapolis, Indiana
  - LSU Health Sciences Center - Shreveport, Shreveport, Louisiana
  - National Heart Lung and Blood Institute, Bethesda, Maryland
  - Kaiser Permanente - Largo Medical Center, Largo, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Boston Medical Center & Boston University School of Medicine, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Southern Specialty Clinic, Flowood, Mississippi
  - Mississippi Center for Advanced Medicine, Madison, Mississippi
  - Cure 4 The Kids Foundation, A Division of Roseman University of Health Sciences, Las Vegas, Nevada
  - East Carolina University - Brody School of Medicine, Greenville, North Carolina
  - Penn Medicine - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Lifespan at Rhode Island Hospital, Providence, Rhode Island
  - University of Texas Health Science Center of Houston, Houston, Texas
  - Texas Children's Hospital, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Seattle Cancer Care Alliance, University of Washington, Seattle, Washington
- Belgium (5):
  - Hôpital Erasme, Anderlecht, Brussels Capital
  - Universitair Ziekenhuis Antwerpen, Edegem, Brussels Capital
  - ZAS Cadix, Antwerp
  - CHR de la Citadelle, Liège
  - Clinique CHC MontLégia, Liège
- Brazil (8):
  - Multihemo Servicos Medicos S/A, Recife, Pernambuco
  - Hospital de Clinicas de Porto Alegre (HCPA) - PPDS, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas Da Pontificia Universidade Catolica Do Rio Grande Do Sul (PUCRS), Porto Alegre, Rio Grande do Sul
  - Hospital de Clínicas da Unicamp, Campinas, São Paulo
  - Hospital Das Clínicas da Faculdade de Medicina de Ribeirão Preto - USP, Ribeirão Preto, São Paulo
  - Praxis Pesquisa Medica, Santo André, São Paulo
  - HEMORIO Instituto Nacional de Hematologia, Rio de Janeiro
  - Hospital das Clínicas da Faculdade de Medicina da Universidad de São Paulo, São Paulo
- Canada (4):
  - McMaster University - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - University Health Network, Toronto, Ontario
  - CHU Montreal, Montreal, Quebec
  - McGill University Health Center, Montreal, Quebec
- France (6):
  - Hopitaux de La Timone, Marseille, Bouches-du-Rhône
  - Hôpital Pellegrin, CHU de Bordeaux, Bordeaux, Gironde
  - CHU Guadeloupe, Pointe à Pitre, Guadeloupe
  - Institut Universitaire du Cancer de Toulouse - Oncopole, Toulouse, Haute-Garonne
  - CHU Hôpital Henri Mondor, Créteil, Val-de-Marne
  - Hôpital Européen Georges Pompidou, Paris, Île-de-France Region
- Germany (2):
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Regensburg, Regensburg
- Israel (3):
  - HaEmek Medical Center, Afula
  - Rambam Medical Center, Haifa, Ḥeifā
  - Ziv Medical Center, Safed, Ḥeifā
- Italy (6):
  - A.O.R.N. "A. Cardarelli", Napoli, Campania
  - AOU dell'Università degli Studi della Campania Luigi Vanvitelli, Napoli, Campania
  - Azienda Ospedaliero Universitaria Di Modena Policlinico, Modena, Emilia-Romagna
  - IRCCS Ospedale Pediatrico Bambino Gesù - INCIPIT - PIN, Rome, Lazio
  - Ente Ospedaliero Ospedali Galliera, Genoa, Liguria
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia-Cervello, Palermo, Sicily
- Kenya (7):
  - Kemri Usamru, Kisumu, Western
  - Kondele Children's Hospital, Kisumu
  - Victoria Biomedical Research Institute (VIBRI), Kisumu
  - KEMRI CRDR Clinical Research Clinic Nairobi, Nairobi
  - KEMRI/CRDR Siaya Clinical Research Annex, Nairobi
  - Strathmore University, Nairobi
  - Gertrude's Children's Hospital, Nairobi
- Lebanon (4):
  - American University of Beirut Medical Center, Beirut, Beyrouth
  - Nini Hospital, Tarablus, Mohafazat Liban-Nord
  - American University of Beirut Medical Center, Beirut
  - Hammoud Hospital University Medical Center, Sidon
- Netherlands (2):
  - Erasmus MC, Rotterdam, South Holland
  - Universitair Medisch Centrum Utrecht, Utrecht
- Nigeria (3):
  - National Hospital Abuja, Abuja, Federal Capital Territory
  - University of Abuja Teaching Hospital, Abuja, Federal Capital Territory
  - Lagos University Teaching Hospital, Surulere, Lagos
- Sultan Qaboos University Hospital, Hematology Department, COM&HS, Muscat, Musqal, Oman
- Saudi Arabia (2):
  - King Khalid University Hospital, Riyadh, Ar Riya
  - King Abdullah International Medical Research Center, Riyadh
- Turkey (Türkiye) (2):
  - Hacettepe University, Ankara, Adana
  - Acibadem Adana Hospital, Seyhan, Adana
- United Kingdom (7):
  - Evelina Children's Hospital, London, City of London
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Guy's and St Thomas' NHS Foundation Trust, London
  - King's College Hospital NHS Foundation Trust, London
  - Hammersmith Hospital, London
  - University College London Hospitals (UCLH), London
  - Manchester Royal Infirmary, Manchester University NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Idowu M, Otieno L, Dumitriu B, Lobo CLC, Thein SL, Andemariam B, Nnodu OE, Inati A, Glaros AK, Bartolucci P, Colombatti R, Taher AT, Abboud MR, Darbari D, Ataga KI, Antmen AB, Kuo KHM, de Souza Medina S, Oluyadi A, Iyer V, Morris S, Yates AM, Shao H, Patil S, Urbstonaitis R, Zaidi AU, Gheuens S, Smith WR. Safety and efficacy of mitapivat in sickle cell disease (RISE UP): results from the phase 2 portion of a global, double-blind, randomised, placebo-controlled trial. Lancet Haematol. 2025 Jan;12(1):e35-e44. doi: 10.1016/S2352-3026(24)00319-3. Epub 2024 Dec 4. PMID 39644907
- [Derived] van Dijk MJ, Rab MAE, van Oirschot BA, Bos J, Derichs C, Rijneveld AW, Cnossen MH, Nur E, Biemond BJ, Bartels M, Jans JJM, van Solinge WW, Schutgens REG, van Wijk R, van Beers EJ. One-year safety and efficacy of mitapivat in sickle cell disease: follow-up results of a phase 2, open-label study. Blood Adv. 2023 Dec 26;7(24):7539-7550. doi: 10.1182/bloodadvances.2023011477. PMID 37934880
- [Derived] Obadina M, Wilson S, Derebail VK, Little J. Emerging Therapies and Advances in Sickle Cell Disease with a Focus on Renal Manifestations. Kidney360. 2023 Jul 1;4(7):997-1005. doi: 10.34067/KID.0000000000000162. Epub 2023 May 31. PMID 37254256